CLINICAL TRIAL: NCT05440071
Title: PoSt-market Assessment on Safety and Performance of J-sHAPed xFINE Lead
Acronym: SHAPE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Other Study IDs: LXFP01 - SHAPE
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: JX- XFINE lead — Pacemaker subjects implanted with one JX - XFINE passive pacing lead

SUMMARY:
The primary objective of this study is to evaluate the safety and the electrical performances of the right atrial J-shape (JX model) XFINE endovascular passive lead at 3 months post implant.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has reviewed, signed and dated the informed consent form
2. Subject newly implanted (de novo) with a JX XFINE within 10 days, connected to a dual chamber (DR) pacemaker from MicroPort CRM S.r.l and any commercially available IS-1 right ventricular lead
3. Subject is willing and capable of participating in all testing/ visits associated with this clinical study at an approved clinical study center and at the intervals defined by this protocol.

Exclusion Criteria:

1. Subjects with documented permanent or persistent AF
2. Included in another clinical study that could confound the results of this study such as studies involving intra-cardiac device
3. Subject has had any pacing or ICD system implants
4. Patient implanted despite a contraindication for cardiac pacing system implantation (i.e. patient implanted with a defibrillator, patient contraindicated for a single dose of 310 μg of dexamethasone sodium phosphate, patient implanted with a tricuspid replacement heart valve or with a significant tricuspid valve disease that may lead to future replacement heart valve surgery)
5. Age less than 18 years old, incapacitated or under guardianship or kept in detention
6. Life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject indicated for a de novo implantation of a dual chamber (DR) pacemaker as per Guidelines on cardiac pacing and cardiac resynchronization therapy.
Sampling Method: Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Safety of the right atrial J-shape (JX model) XFINE endovascular passive lead at 3 months post implant. | 3 months
Electrical performances of the right atrial J-shape (JX model) XFINE endovascular at 3 months | 3 months